CLINICAL TRIAL: NCT02489409
Title: EndostarTM Injection Combined With Gemcitabine+Platinum (GP)/Navelbine+Platinum (NP)/Gemcitabine+Xeloda (GX)/Navelbine+Xeloda (NX) in Treatment of Recurrent Metastatic Breast Cancer: A Randomized, Opened and Controlled Clinical Study
Brief Title: Recombinant Human Endostatin (EndostarTM) Injection in Treatment of Recurrent Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Shun-E Yang, Asistant investiagtor, clinical research, Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XinjiangMU001
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Endostatins; Gemcitabine; Vinorelbine; Platinum; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Gemcitabine (Gem): 1.0 m/m2, iv 0.5h, d1, 8; Navelbine (NVB): 40 mg/d, iv, d1, 8; Platinum (DDP): 30 mg/m2, iv 3h, d1-3; Xeloda Tablets: 2 000 mg/m2, po, d1-14; EndostarTM Injection: 210 mg in 279 mL normal saline (NS), continuous pump, d1-d10 (2.5 mL/h).
  Interventions: Drug: EndostarTM Injection; Drug: Gemcitabine; Drug: Navelbine; Drug: Platinum; Drug: Xeloda Tablets:
- Control group (Active Comparator): Gemcitabine (Gem): 1.0 m/m2, iv 0.5h, d1, 8; Navelbine (NVB): 40 mg/d, iv, d1, 8; Platinum (DDP): 30 mg/m2, iv 3h, d1-3; Xeloda Tablets: 2 000 mg/m2, po, d1-14.
  Interventions: Drug: Gemcitabine; Drug: Navelbine; Drug: Platinum; Drug: Xeloda Tablets:

INTERVENTIONS:
Drug: EndostarTM Injection — 210 mg in 279 mL normal saline (NS), continuous pump, d1-d10 (2.5 mL/h)
  Other Names: Endostatin
  Arms: Experimental group
Drug: Gemcitabine — 1.0 m/m2, iv 0.5h, d1, 8
  Other Names: GEM
Drug: Navelbine — 40 mg/d, iv, d1, 8
  Other Names: NVB
Drug: Platinum — 30 mg/m2, iv 3h, d1-3
  Other Names: DDP
Drug: Xeloda Tablets: — 2 000 mg/m2, po, d1-14
  Other Names: ECX

SUMMARY:
Endostatin has been widely applied for the clinical treatment of partial primary and metastatic solid tumors. Endostatin combined with chemotherapy has achieved favorable progression in the treatment of non-small cell lung cancer (NSCLC). However, the research about the efficacy of Endostatin on breast cancer has just started. Breast cancer is a highly-differentiated solid tumor, indicating that it is also an indicator for Endostatin therapy. Additionally, after chemo- and radiotherapy, the primary nidi of patients with advanced breast cancer may also lead to rapid development of tumors in other locations. So Endostatin combined with chemotherapy can also improve the prognosis of patients with recurrent metastatic breast cancer, but there is rare any report at home and abroad. To further explore the above research, this study designed a randomized, opened and controlled clinical study to observe the clinical efficacy of EndostarTM Injection combined with GP/NP/GX/NX in the treatment of recurrent metastatic breast cancer.

DETAILED DESCRIPTION:
Large amounts of studies have proved that the development of tumor vessels mainly depend on the activation, proliferation, adhesion and maturity of vascular endothelial cells, which may also become the targets of vascular inhibitors. At present, Avastin, an anti-angiogenesis drug, has been marketed in Euopean and American countries, and another 30 kinds of vascular inhibitors are still in trails. Endostatin has been widely applied for the clinical treatment of partial primary and metastatic solid tumors. Endostatin combined with chemotherapy has achieved favorable progression in the treatment of non-small cell lung cancer (NSCLC). However, the research about the efficacy of Endostatin on breast cancer has just started. Breast cancer is a highly-differentiated solid tumor, indicating that it is also an indicator for Endostatin therapy. Additionally, after chemo- and radiotherapy, the primary nidi of patients with advanced breast cancer may also lead to rapid development of tumors in other locations. So Endostatin combined with chemotherapy can also improve the prognosis of patients with recurrent metastatic breast cancer, but there is rare any report at home and abroad. To further explore the above research, this study designed a randomized, opened and controlled clinical study to observe the clinical efficacy of EndostarTM Injection combined with GP/NP/GX/NX in the treatment of recurrent metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18～70 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0～1 score;
* All patients were diagnosed as recurrent metastatic breast cancer retreatment by histopathology and computed tomography (CT) examination;
* The measurable nidus≥1: Patients whose nidus diameter ≥ 20 mm by normal CT or magnetic resonance image (MRI) scanning, and ≥ 10 mm by spiral CT scanning;
* Patients whose blood routine, hepatorenal function, electrolyte and cardiac function were basically normal without dysfunction of primary organs. White blood cell count (WBC) ≥4.0×109/L, neutrophile granulocyte count ≥1.5×109/L, platelet (PLT) count ≥100×109/L, hemoglobin (HGB) ≥95 g/L, serum bilirubin (BIL) ≤1.5-fold upper limit of normal value, alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤2-fold upper limit of normal value, and serum creatinine (Scr) ≤1.5mg/dl;
* The expected survival time >3 months;
* Patients who could understand this study status and had signed the informed consent forms.

Exclusion Criteria:

* Patients who had history of allergic responses to biological agents;
* Patients who were receiving other anti-tumor therapies;
* Patients without measureable nidus;
* Others, including one of the following conditions: patients with uncontrolled central nervous system (CNS) metastatic nidi, with dysfunction of important organs and severe cardiac diseases (congestive heart failure, uncontrollable arrhythmia, and angina pectoris, valvular heart disease, myocardial infarction and refractory hypertension that required long-term drug administration), with chronic infectious wound and with history of uncontrollable psychosis, and women in pregnant or lactation period.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
response rate | 2 years
  response rate that defined as the total ratio of study subjects with complete response, complete response unconfirmed and partial response after treatment. ORR=(CR+ CRu+ PR)cases/total cases×100%.

SECONDARY OUTCOMES:
clinical benefit rate | 2 years
  clinical benefit rate that defined as the total ratio of study subjects with complete response，partial response and stable disease more than 24 months after treatment.
progression-free survival | 2 years
  Progression-free survival (PFS) defined as the ratio of study subjects who had disease progression or died from the start of randomization.
median survival time | 2 years
  median survival time defined as the corresponding survival time when the cumulative survival rate is 50%.
overall survival | 2 years
  overall survival rate (OS) that defined as the ratio of study subjects who survived after randomization
adverse responses | 2 years
  adverse responses that defined as the evaluated by rates of all adverse reactions caused by Recombinant Human Endostatin and the changes of all indexes before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shun-E Yang, Professor, Principal Investigator — Third Affiliated Hospital of Xinjiang Medical University
Locations (1):
- Third Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No